CLINICAL TRIAL: NCT02234518
Title: Evaluation of Changes in Gut Transit Time and Gastrointestinal Symptoms Following the Consumption of a Fiber Containing Product in Adults With Constipation
Brief Title: Fibers and Gut Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 12.04.NRC
Record Dates: First submitted 2014-09-02; First posted 2014-09-09 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-11

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- High quantity fiber food product (Experimental)
  Interventions: Other: High quantity fiber
- Low quantity fiber food product (Experimental)
  Interventions: Other: Low quantity fiber
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Other: High quantity fiber — The intervention type is food product
  Arms: High quantity fiber food product
Other: Low quantity fiber — The intervention type is food product
  Arms: Low quantity fiber food product
Other: Placebo
  Arms: Placebo

SUMMARY:
Gastrointestinal discomfort regularly affects >25% of the population worldwide. One of the major contributors to GI discomfort is constipation, which has a prevalence of ~15% and symptoms of which have a significant negative impact on the sufferer's quality of life. One of the hallmarks of chronic constipation is slow progression of contents through the gut (i.e. slow gut / colonic transit time), which may be associated with hard stools that are difficult to expel.

Dietary fiber supplements are widely used as a first-line treatment for constipation although little Level 1 evidence exists to support its use in adults. The effectiveness of different fiber supplements is difficult to compare given wide differences in water-retention capabilities and effects on the colonic microbial ecology. Given the promising, yet largely unsubstantiated, benefits of fiber supplementation on symptoms of functional constipation, the objective of this clinical trial is to evaluate tolerance and effectiveness of four week supplementation of a fiber product, in a dose-ranging fashion, on whole gut transit time and gastrointestinal symptoms in adults with functional constipation.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 18-75; female subjects of child-bearing potential must be willing to use a reliable method of contraception throughout the study period
* BMI: 18.5 - 29.9 kg/m2
* Recruitment based on simplified core ROME III diagnostic criteria for functional constipation (based on specific screening questions):a). average Bristol stool type of 1 - 4 AND frequency of 1 - 3 spontaneous bowel movements (SBMs) per week b). plus at least ONE of: straining on at least 25% of defaecations; sensation of incomplete evacuation on at least 25% of defaecations; sensation of anorectal obstruction / blockage on at least 25% of defaecations; use of manual manoeuvres on at least 25% of defaecations
* Cleveland Clinic constipation score (CCCS) of 8-20
* Low-moderate fiber intake (≤18g) determined by the semi-quantitative food intake screener known as the Block Fiber Screener
* Ability to understand the patient information sheet and instructions in Dutch, and able to provide informed consent

Exclusion Criteria:

* Subjects who report lactose intolerance and/or are allergic to soy or cow milk protein
* Pregnant or breast-feeding women
* Ongoing other diagnosed gastrointestinal disease or complication (Crohn's disease, Coeliac disease, chronic diarrhoea)
* Any clinical relevant abnormalities in the screening visit medical examination or alarm features such as sudden unintentional weight loss, rectal bleeding, recent change in bowel habit (<3 months), abdominal pain and stool positive for occult blood
* Prior abdominal surgery (including gastric bypass or laparoscopic banding), except cholecystectomy and appendicectomy
* Neurologic diseases such as multiple sclerosis, stroke, spinal cord injury, Hirschsprung disease
* Chronic medication that in opinion of the investigator would impact gut motility
* Illness that may preclude the subject's ability to complete the study or that may confound the study outcomes (e.g. bowel cancer, prostate cancer, terminal illness, severe cardiovascular disease, chronic renal failure or eating disorders) or any other serious illness resulting in >2 weeks inability to work in the 3 months before the study start
* Subjects with co-morbid illnesses such as cardiovascular, endocrine, renal or other chronic disease likely to affect gut motility or limit normal functions (e.g. reduced mobility or increased fragility)
* Ongoing alcohol, drug, or medication abuse (anamnesis only)
* Self-reported symptoms of pelvic organ prolapse
* Moderate or severe active local anorectal problems such as recurrent anal fissures, bleeding, large prolapsing haemorrhoids
* Regular use of fiber supplementation (e.g. Fybogel, Lactulose) (i.e. no more than 1 standard dose) over the week prior to the screening visit and no more than 6 standard doses in the past 1 month prior to the screening visit
* Participation in another study with any investigational product within 3 months of screening
* Investigator believes that the participant is physically or mentally unfit to participate in the trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Whole gut transit time | After 2 weeks consumption of the study product
  To evaluate change in whole gut transit time 2 weeks after consumption of the study product in constipated patients consuming the study product containing fiber in high quantity, compared to those consuming placebo

SECONDARY OUTCOMES:
Gastrointestinal symptoms | After 2&4 weeks consumption of the study product
  To evaluate change in Gastrointestinal symptoms 2&4 weeks after consumption of the study product in all groups
Regional colonic transit time | After 2 weeks consumption of the study product
  To evaluate change in the regional (right colon, left colon, and rectosigmoid tranist time 2 weeks after consumption of the study product in all groups
Whole gut transit time | After 2 weeks consumption of the study product
  To evaluate change in whole gut transit time 2 weeks after consumption of the study product in constipated patients consuming the study product containing fiber in low quantity, compared to those consuming placebo
Tolerance | After 1&2&4 weeks consumption of the study product
  To assess tolerance to the study product 1&2&4 weeks after consumption in all groups, using a questionnaire

OTHER OUTCOMES:
Adverse Events | Through the study product consumption period (4 weeks)
  Adverse events assessed as treatment emergent adverse events (TEAEs)
Gut Health Insight Survey | At screening, after informed consent
  To gain insights into patient-specific constipation symptomology

CONTACTS AND LOCATIONS:
Overall Officials: Diederick E. Grobbee, Prof, MD, PhD, Principal Investigator — Julius Clinical
Locations (1):
- Julius Clinical, Zeist, Netherlands